CLINICAL TRIAL: NCT00143078
Title: The Effects of Morbid Obesity and Weight Loss on Reproductive Function: The Bariatric Surgery Model
Brief Title: Obesity and Weight Loss on Reproductive Function
Status: Terminated | Type: Observational
Why Stopped: Close-out of the grant - study ceased on 1/1/2010
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Tobacco Settlement Grant (Unknown)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Other Study IDs: 19366
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: Obesity; Reproduction; Weight Loss; Reproductive System
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood & urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine how obesity and weight loss following bariatric surgery affect reproductive function. The study is particularly interested in how changes in hormones (those produced in the stomach and fat tissue) following weight loss affect reproductive function. Specifically, we, the researchers at Penn State University, propose to characterize reproductive abnormalities in morbidly obese men and women. We hypothesize that morbid obesity leads to reproductive abnormalities in men and women. We plan to examine the short-term effects of alteration in GI hormones after bariatric surgery on reproductive function. We hypothesize that bariatric surgery radically alters GI hormone expression, resulting in immediate changes to the hypothalamic-pituitary-gonadal axis in men and women. Lastly, we, the researchers, plan to examine the long-term effects of weight loss and changes in adipokines on reproductive function. We hypothesize that the changes in adipokine levels resulting from fat mass reduction lead to substantial long-term improvements in reproductive function and fertility. We also hypothesize that there are sexual dimorphisms in adipokine levels following weight loss, with women experiencing larger changes than men.

DETAILED DESCRIPTION:
Obesity may influence female reproduction through a variety of mechanisms including: suppressing ovulation; inhibiting ovarian follicular development; and altering endometrial development and implantation. In males, obesity may impair reproductive function by several mechanisms including: decreasing libido, causing erectile dysfunction, influencing semen composition, or sperm function. Therefore the long term goal of the current project is to understand the impact of severe obesity on reproductive function and how this is influenced by dramatic weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of greater than 40 or a BMI between 35.5-39.9 and has a weight related health problem, such as diabetes or high blood pressure.
* Failed medical weight loss
* Ages of 18-40
* Not using hormonal contraception or sex steroids
* Subject is premenopausal and has not undergone a bilateral oophorectomy or hysterectomy
* Subject's obesity has no medical explanation (hypothyroidism, Cushing's Syndrome, genetic)

Exclusion Criteria:

* Not willing to make a lifelong commitment to the diet and exercise guidelines following bariatric surgery
* Subject is pregnant or lactating
* Not willing to use barrier contraceptives or intrauterine device (IUD) to prevent pregnancy for one year following bariatric surgery
* Post-menopausal, either surgical or natural
* Subject has had a vasectomy
* Subject is a smoker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants eligible for bariatric surgery; BMI >40 or between 35 and 39.9 with a weight related health problem; Failed medical weight loss; Ages 18-40; Not using hormonal contraceptives; Females have not undergone and bilateral oophrectomy or hysterectomy; Males have not had a vasectomy
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Integrated levels of urinary progestin (Pregnanediol-3-Glururonide or Pd3G) at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Legro, M.D., Principal Investigator — Penn State University/Milton S. Hershey Medical Center
Locations (1):
- The Penn State Hershey Medical Center, Hershey, Pennsylvania, United States